CLINICAL TRIAL: NCT06825702
Title: A Phase 2, Open-label, Multiple Dose Study of the Safety, Tolerability and Efficacy of Intravitreal KIO-104 in Patients With Macular Edema (KLARITY-1)
Brief Title: Safety, Tolerability and Efficacy of Intravitreal KIO-104 in Patients With Macular Edema
Acronym: KLARITY-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kiora Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KIO-104-2100
Record Dates: First submitted 2025-02-04; First posted 2025-02-13 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-07

CONDITIONS: Macular Edema
Keywords: Macular Edema
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Dose KIO-104: 2-weekly (Experimental): 2-weekly dosing
  Interventions: Drug: KIO-104
- High Dose KIO-104: 2-weekly (Experimental): 2-weekly dosing
  Interventions: Drug: KIO-104
- Low or High Dose KIO-104: 2-weekly (Experimental): 2-weekly dosing
  Interventions: Drug: KIO-104
- Low or High Dose KIO-104: 4-weekly (Experimental): 4-weekly dosing
  Interventions: Drug: KIO-104

INTERVENTIONS:
Drug: KIO-104 — KIO-104 is an ophthalmic formulation for IVT injection of the active pharmaceutical ingredient (API) KIO-100, a novel, non-steroidal, small molecule inhibitor of dihydroorotate dehydrogenase (DHODH).

SUMMARY:
This is a multi-center, open label study to assess the safety, tolerability, and efficacy of KIO-104 administered by IVT injection to the study eye of eligible participants with macular edema.

DETAILED DESCRIPTION:
In Part A of the study, the safety and efficacy of up to three doses (administrations) of KIO-104, administered every 2 weeks, will be investigated in 2 possible dose cohorts.

Cohort 1: Low dose KIO-104 administered to the study eye Cohort 2: High dose KIO-104 administered to the study eye Part B of the study will investigate the safety and efficacy of up to three doses (administrations) of KIO-104 with 2 different dosing regimens (every 2 weeks or every 4 weeks), in participants with macular edema at a dose selected from Part A.

Cohort 3A: KIO-104 administered to the study eye every 2 weeks Cohort 3B: KIO-104 administered to the study eye every 4 weeks

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria:

1. Be aged 18 to 85 years inclusive at the time of consent.
2. Provide informed consent prior to any study procedures, as stipulated by local laws, Ethics Committee (EC) and Regulatory Authority (RA) guidelines.
3. Be willing and able to follow all study instructions, attend all study visits, and complete all study assessments.
4. Have a clinical diagnosis of ME in the study eye secondary to non-infectious uveitis, retinal vein occlusion, diabetic retinopathy or cataract surgery.
5. If currently receiving systemic corticosteroid therapy or immunosuppressive therapy (or any combination thereof), be on a stable dose of therapy for at least 3 months prior to Screening and during the study.
6. Have a Central Subfield Thickness (CST) of ≥ 350 µm.
7. Have a Best Corrected Visual Acuity (BCVA) in the study eye of:

   1. ≤ 20/32 (Feet); logMAR ≥ 0.2
   2. ≥ 20/800 (Feet); log MAR ≤ 1.6
8. Have media clarity and pupillary dilation sufficient for adequate visualization and assessment of the study eye.
9. Be willing to avoid disallowed medications and treatments for the duration of the study.
10. Agree to follow appropriate contraception requirements from screening until 3 months after the last dose of the study drug.

    1. Participants assigned female at birth who are of child-bearing potential (OCBP) must agree to a pregnancy test at Screening and prior to each dose of investigational medicinal product (IMP) and use an acceptable method of birth control including oral, transdermal, injectable, or implantable hormonal contraception, intrauterine device, abstinence from intercourse with partner assigned male at birth, or surgical sterilisation of partner assigned male at birth.
    2. Participants assigned female at birth are not OCBP if they have had a hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or are post-menopausal by at least 12 months. Post-menopausal status of amenorrheic female participants should be confirmed at Screening through testing of follicle-stimulating hormone (FSH) as per analysing laboratory threshold.
    3. Participants assigned male at birth with a partner OCBP must be surgically sterile for at least 3 months prior to starting study drug, or ensure their partner uses contraception as outlined above, and must use a male condom. Participants assigned male at birth must not donate sperm from Screening until 3 months after the last dose of IMP.
    4. Participants who have practiced true abstinence for at least 1 year due to usual and preferred lifestyle choice are exempt from contraceptive requirements. If a participant who is abstinent becomes sexually active, they must agree to use appropriate contraception as described above.

Exclusion Criteria:

Participants must not meet any of the following criteria:

1. Have media opacities (cornea, anterior or posterior synechia, cataract, vitreous haze and others) of either eye that preclude investigation and documentation of the posterior pole and intravenous fluorescein angiography, or optical coherence tomography evaluation in the study eye.
2. Receive local or systemic biologicals (i.e. tumour necrosis factor [TNF]-blockers, B-cell blockers, cytokines, cytokine-blockers, receptor antagonists) 90 days prior to Day 1 or planned during the study.
3. Receive treatment with cyclophosphamide or chlorambucil during the study.
4. Receive intravitreal injections (including but not limited to anti-vascular endothelial growth factors) 90 days prior to Day 1 or planned during the study.
5. Receive a posterior subtenon's or orbital floor injection of steroids 90 days prior to Day 1 or planned during the study.
6. Have any implantable corticosteroid-eluting device (Ozurdex, Iluvien, Retisert, triamcinolone intravitreal implant, fluocinolone intravitreal implant) in the study eye, with the following exceptions:

   1. If the device had been removed more than 90 days prior to Day 1 of the study.
   2. If Ozurdex® had been implanted at least 6 months before Day 1 of the study.
   3. If Iluvien® or Retisert® had been implanted at least 3 years before Day 1 of the study.
   4. Use of topical steroids are permissible provided the participant is receiving a stable dose for at least 3 months prior to Screening and during the study.
7. Have ocular surgery (including cataract extraction, vitreoretinal or scleral buckling surgery) in the study eye, within 90 days prior to Day 1, or planned during the study.
8. Have a capsulotomy in the study eye, within 30 days prior to Day 1, and during the study.
9. Have Intraocular pressure (IOP) ≥ 25 mmHg in the study eye (glaucoma patients maintained on no more than one topical medication with IOP < 25 mmHg are allowed to participate).
10. Have ocular hypotony (IOP < 6 mmHg).
11. Have aphakia or anterior chamber lens in the study eye.
12. Have visible scleral thinning, scleral ectasia or keratoconus in the study eye.
13. Have presence of any ocular malignancy in either eye.
14. Have evidence of any other clinically significant ocular disease that might interfere with the study assessments.
15. Have ocular or periocular (either eye) or systemic infection and/or a temperature greater than 38.0°C, or the use of systemic or topical ocular antibiotics within 14 days of Day 1.
16. Have a psychiatric condition that, in the investigator's opinion, precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within five years prior to screening, a history of suicide plan.
17. Have any clinically significant abnormality at screening determined by medical and ophthalmic history, vital signs, clinical biochemistry, hematology, urinalysis, or a 12-lead electrocardiogram (ECG), as assessed by the investigator, which might interfere with the study assessments or the ability of the participant to complete the study.
18. Have any other medical condition or significant co-morbidities, or any finding during screening, which in the view of the investigator is likely to interfere with the study or put the participant at risk, confound study data, or interfere significantly with study participation.
19. Have participated in any other investigational drug or device clinical trial within 90 days prior to Day 1 or planning to participate in other investigational drug or device clinical trials during the study and within 90 days following Day 1. This includes both ocular and non-ocular clinical trials.
20. Receive any anticoagulant or thrombocyte aggregation inhibiting agent (marcumar, warfarin, heparin, enoxaparin, apixaban, rivaroxaban, pentosanpolysulfate, dabigatran, aspirin and others) within 14 days prior to Day 1 or planned during the study.
21. Have a known allergy or hypersensitivity to the study medication, any component of the delivery vehicle, any corticosteroids, any diagnostic agents used during the study (e.g., fluorescein, dilation drops), or any other standard of care medications likely to be used during the study (e.g., antibiotic drops, povidone, rescue medications).
22. Be pregnant or breast-feeding, or plan to become pregnant during the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 23months
  The primary objective is safety and tolerability. The incidence of AEs will be presented by System Organ Class (SOC) and Preferred Term (PT) by dose cohorts.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Sydney Eye Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Centre for Eye Research Australia, East Melbourne, Victoria
  - Lions Eye Institute Limited, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thurau S, Deuter CME, Heiligenhaus A, Pleyer U, Van Calster J, Barisani-Asenbauer T, Obermayr F, Sperl S, Seda-Zehetner R, Wildner G. A new small molecule DHODH-inhibitor [KIO-100 (PP-001)] targeting activated T cells for intraocular treatment of uveitis - A phase I clinical trial. Front Med (Lausanne). 2022 Oct 17;9:1023224. doi: 10.3389/fmed.2022.1023224. eCollection 2022. PMID 36325389